CLINICAL TRIAL: NCT04505423
Title: Evaluation of Outcomes Related to Cerebrospinal Fluid Drains Placed Either With or Without Fluoroscopic Guidance for Aortic Surgery
Brief Title: Evaluation of Outcomes Related to Cerebrospinal Fluid Drain Placement
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: UNC Medical Alumni (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-0727
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cerebrospinal Fluid Drainage
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blind CSF Drain Placement — CSF Drain placement without fluoroscopic image guidance.
Procedure: Fluoroscopy-guided Drain Placement — CSF Drain placement utilizing fluoroscopic image guidance.

SUMMARY:
The purpose of this study is to compare the rate and severity of complications associated with CSFD placement either with or without fluoroscopic guidance.

DETAILED DESCRIPTION:
Patients undergoing thoracoabdominal aortic aneurysm (TAAA) repair are at risk of suffering devastating spinal cord injury (SCI), rendering them with a permanent neurologic deficit, paraplegia, or paraparesis. Despite huge success over the last several decades with the introduction of innovative protective maneuvers, such as the use of cerebrospinal fluid drains (CSFDs), the rate of these complications remains around 5%. Spinal cord perfusion can be compromised during aortic surgery and the intrathecal decompression achieved by CSFDs functions to increase the pressure gradient of blood flow, thereby optimizing spinal cord perfusion during aortic surgery. There are two methods commonly used to place cerebrospinal fluid drains: blind placement and with fluoroscopic guidance. Prior to 2016, CSFDs at UNC hospital were primarily placed without image guidance. However, hospital policy then transitioned to having all CSFDs placed using fluoroscopic guidance. To the investigators' knowledge, there are no reported studies directly comparing clinical outcomes of CSFDs placed by these methods. Given the increased cost and radiation exposure associated with the use of fluoroscopy, a better understanding of comparative outcomes has great potential clinical value. Therefore, the investigators propose to compare the rate and severity of complications associated with CSFD placement either with or without fluoroscopic guidance.

ELIGIBILITY:
Inclusion Criteria:

* CSF drain placed from 2010 to present prior to undergoing aortic surgery

Exclusion Criteria:

* Patients under 18 years of age
* Patients undergoing emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UNC Hospital System Patients
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Rate and Severity of Complications Related Associated with CSFD placement | From admission to discharge, up to 2 weeks
  The rate and severity of complications associated with CSFD placement with or without fluoroscopic guidance via a chart review. This will be assessed using quantitative methods such as vital signs and lab-work drawn relating to the procedure as well as qualitative variables through clinical notes.

CONTACTS AND LOCATIONS:
Overall Officials: Harendra Arora, MD, MBA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Data will be shared beginning 9 to 36 months following publication.
Access Criteria: Data will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Svensson LG, Crawford ES, Hess KR, Coselli JS, Safi HJ. Experience with 1509 patients undergoing thoracoabdominal aortic operations. J Vasc Surg. 1993 Feb;17(2):357-68; discussion 368-70. PMID 8433431
- [Background] Safi HJ, Estrera AL, Miller CC, Huynh TT, Porat EE, Azizzadeh A, Meada R, Goodrick JS. Evolution of risk for neurologic deficit after descending and thoracoabdominal aortic repair. Ann Thorac Surg. 2005 Dec;80(6):2173-9; discussion 2179. doi: 10.1016/j.athoracsur.2005.05.060. PMID 16305866